CLINICAL TRIAL: NCT02080130
Title: Efficacy of Two Probiotic Preparations in Children With Acute Viral Diarrhoea, Randomised Controlled Trial
Brief Title: Efficacy of Two Probiotic Preparations in Children With Acute Diarrhoea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants.
Sponsor: Sinaloa Pediatric Hospital (Other)
Responsible Party: Principal Investigator, Giordano Perez Gaxiola, Pediatrician, Sinaloa Pediatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HPS-03
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Gastroenteritis
Keywords: Gastroenteritis; diarrhea
MeSH Terms: conditions — Gastroenteritis; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saccharomyces boulardii (Experimental): FLORATIL®. Saccharomyces boulardii 200 mg sachet. One sachet orally, BID, for 5 days.
  Interventions: Dietary Supplement: Saccharomyces boulardii
- Probiotics combination (Experimental): LACTIPAN®. Probiotics combination sachet. One sachet orally, BID, for 5 days. Lactobacillus acidophilus............. 1.00 x 109 cfu Lactobacillus casei........................ 1.00 x 109 cfu Lactobacillus rhamnosus............. 4.40 x 108 cfu Lactobacillus plantarum............... 1.76 x 108 cfu Bifidobacterium infantis................ 2.76 x 107 cfu Streptococcus thermophillus....... 6.66 x 105 cfu
  Interventions: Dietary Supplement: Probiotics combination
- Placebo (Placebo Comparator): Placebo sachet. One sachet orally, BID, for 5 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Saccharomyces boulardii — FLORATIL®. Saccharomyces boulardii 200 mg sachet. One sachet orally, BID, for 5 days.
  Arms: Saccharomyces boulardii
Dietary Supplement: Probiotics combination — LACTIPAN®. Probiotics combination sachet. One sachet orally, BID, for 5 days. Lactobacillus acidophilus............. 1.00 x 109 cfu Lactobacillus casei........................ 1.00 x 109 cfu Lactobacillus rhamnosus............. 4.40 x 108 cfu Lactobacillus plantarum............... 1.76 x 108 cfu Bifidobacterium infantis................ 2.76 x 107 cfu Streptococcus thermophillus....... 6.66 x 105 cfu
  Arms: Probiotics combination
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine which of two different preparations of probiotics is effective in the treatment of acute viral diarrhoea in children.

DETAILED DESCRIPTION:
Children and infants, aged 1 month to 5 years, with acute diarrhoea, will be randomised to receive either saccharomyces boulardii, a combination probiotic (Lactobacillus acidophilus, Lactobacillus casei, Lactobacillus rhamnosus, Lactobacillus plantarum, Bifidobacterium infantis, Streptococcus thermophillus) or placebo, to determine if one shortens the duration of diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute viral gastroenteritis

Exclusion Criteria:

* Moderate or severe dehydration
* Malnutrition
* Immunodeficiencies
* Sepsis or bacterial infection
* Previous use of antibiotics, antidiarrheal drugs, or probiotics, in the last four weeks.
* Hospitalisation
* No phone number
* Illiteracy

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Duration of diarrhoea in hours | Up to 7 days

SECONDARY OUTCOMES:
Percentage of children requiring hospitalisation | Up to 7 days
Adverse effects | Up to 7 days
Number of liquid stools | Up to seven days

CONTACTS AND LOCATIONS:
Overall Officials: Giordano Pérez-Gaxiola, MD, Study Chair — Sinaloa Pediatric Hospital
Locations (1):
- Sinaloa Pediatric Hospital, Culiacán, Sinaloa, Mexico